CLINICAL TRIAL: NCT01477294
Title: Effects of Caffeine Ingestion in Total-body Water, Extra and Intracellular Water Distribution, and Energy Metabolism
Brief Title: Effects of Caffeine in Hydration and Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Lisbon (Other)
Responsible Party: Principal Investigator, Analiza M Silva, PhD, Principal Investigator, Technical University of Lisbon
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IHS-2010
Record Dates: First submitted 2011-11-11; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Caffeine
Keywords: Total; Intra and Extracellular Water; Energy Expenditure, Physical Activity; Body Composition; Dilution Techniques
MeSH Terms: conditions — Motor Activity | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine (Experimental): Intervention with Caffeine in a random order
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): Placebo (malt dextrin) administered in a random order
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine — 5 mg/ kg of body weight (capsules), twice a day (morning and afternoon), during 4 days.
  Arms: Caffeine
Drug: Placebo — Malt dextrin (5 mg/kg body mass) twice a day during 4 days
  Arms: Placebo

SUMMARY:
The main purposes of this randomized cross-over trial are to characterize and compare the effects of a moderate dose of caffeine intake in healthy physically active males on hydration and energy metabolism specifically:

1. Total body water and its compartments (intracellular and extracellular) assessed by by dilution techniques, and hydration state by urine specific gravity;
2. Total energy expenditure by double labeled water, resting energy expenditure by indirect calorimetry, and physical activity energy expenditure;
3. Energy expenditure in physical activity of daily living, in particular duration and intensity of activity.
4. If the changes occurred between placebo and caffeine ingestion on the main outcomes were dependent on specific covariates, namely body composition and dietary intake.

DETAILED DESCRIPTION:
Although the effect of caffeine on hydration status, usually assessed by a urine specific gravity test (USG) has been extensively studied no research has been conducted to analyze its effects on total body water and its compartments using reference methods. In addition some uncertainty still remains about the influence of caffeine ingestion on hydration due to methodological limitations, specifically the use of less valid techniques for total-body water assessment, small sample size, and the lack of control for potential confounding factors. The information above specifically the methodological gaps mentioned and an inadequate experimental design lead us to further understand the effect of a moderate dose of caffeine in total body water (TBW) and its intra (ICW) and extracellular (ECW) compartments in non-caffeine consumers during a short-term period (4 days). Additionally, though caffeine effects on energy expenditure has been studied, its influence on physical activity (PA) during free-living conditions using gold standard and objective measures of PA is limited. Therefore, we also investigated the impact of a moderate dose of caffeine on resting energy expenditure (REE), PA energy expenditure (PAEE), total energy expenditure (TEE), and daily time spent in sedentary (DTSS), light (DTSL), moderate (DTSM), and vigorous (DTSV) intensity activities in non-obese physically active males. To overcome the methodological gaps in previous studies we assessed dietary intake and objective measures of physical activity throughout the experimental trial to assure that the same diet and physical activity patterns were maintained. Also it was analyzed if the effect of caffeine was independent of body composition, assessed by dual-energy x-ray absorptiometry.

To perform this research study, a total of 30 non-smoker males, low caffeine users (<100 mg/day), aged 20-39 yrs [body mass (BM): 72.7 ± 8.8 kg; Height: 1.77 ± 0.07 m] were followed in a double-blind crossover experimental design with two conditions in a random sequence: caffeine (5 mg per kg of BM/day) and malt-dextrine as placebo, both through capsules. Conditions lasted for 4 days with a 3-day washout period.

Evaluations were performed at baseline (visit-1), end of condition 1 (visit-2), and end of condition 2 (visit-3). Fat and fat-free masses (FFM) were assessed by dual energy x-ray absorptiometry. TBW and ECW were determined by dilution techniques (deuterium and bromide, specifically) while ICW was calculated as the difference between TBW and ECW (Schoeller et al., 1980. Total body water measurement in humans with 18O and 2H labeled water. Am J Clin Nutr 33:2686-2693). TEE was assessed using doubly labeled water technique by administrating two stable isotopes 2H (deuterium) and 18O (oxygen 18) with a respective dose of 0.1 g / kg and 1.8 g / kg of body water (Schoeller DA, van Santen E, 1982. Measurement of energy expenditure in humans by doubly labeled water method. J Appl Physiol 53:955-959). REE was assessed by indirect calorimetry and PAEE calculated as [TEE-(REE+0.1TEE)]. An accelerometer (ActiGraph, GT1M model, Fort Walton Beach, Florida) was used to estimate DTSS, DTSL, DTSM, and DTSV. The cutoff values used to define the intensity of physical activity and therefore to quantify the mean time in each intensity (sedentary, light, moderate or vigorous) for persons aged 18 years or older were: sedentary: < 100 counts/min; light: 100-2019 counts/min; moderate: 2,020-5,998 counts/min (corresponding to 3-5.9 METs); vigorous: ≥ 5999 counts/min (corresponding to ≥ 6 METs) (Troiano et al. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008;40:181-8).

ELIGIBILITY:
Inclusion Criteria:

* male
* aged 18-39 years old
* body mass index between 18.5 and 29.9 kg/m2
* Subjects had to be free of any major disease with a general healthy status warranted

Exclusion Criteria:

* Smokers
* taking medication or dietary supplements that may interfere with hydration status
* body composition or energy expenditure regulation
* Caffeine consumption > 100 mg/day

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Changes in Total body water (TBW), extracellular water (ECW), intracellular water (ICW), and hydration status from baseline to each experimental condition (Placebo or Caffeine) | day 0, day 4, and day 11
  TBW was assessed by deuterium dilution using a stable Hydra gas isotope ratio mass spectrometer (PDZ, Europa Scientific, Crewe, United Kingdom).ECW was assessed by the sodium bromide dilution method. ICW was calculated as the difference between TBW and ECW. Hydration status was determined based on urine specific gravity (USG) measured by a refractrometer (Urisys 1100 Urine Analyzer, Roche, Portugal)
Changes in total energy expenditure (TEE), resting energy expenditure (REE), and physical activity energy expenditure (PAEE) between each experimental conditions (placebo or caffeine) | Day 4 and day 11
  TEE was assessed by the double labeled water technique, REE by indirect calorimetry, and PAEE calculated as PAEE= TEE - (0.1xTEE + REE), assuming that 10% of TEE is due to the thermogenic effect of food
Changes in daily time spent in sedentary activities (DTSS), light activities (DTSL), moderate activities (DTSM), and vigorous activities (DTSV) between each experimental conditions (placebo or caffeine) | day 4 and day 11
  DTSS, DTSL, DTSM, and DTCV were assessed by accelerometry using cut-off values based on specific counts/min interval

SECONDARY OUTCOMES:
Changes in body composition from baseline to each condition (Placebo or Caffeine) | day 0, day 4, and day 11
  Body composition was assessed by dual energy x-ray absorptiometry (DXA)
Changes in dietary intake (energy and macro nutrient) between each condition (placebo and caffeine) | Day 4 and day 11
  Dietary intake was assessed using a 24-h dietary records.

CONTACTS AND LOCATIONS:
Overall Officials: Analiza M Silva, PhD, Principal Investigator — Faculty of Human Kinetics, Technical University of Lisbon
Locations (1):
- Faculty of Human Kinetics, Lisbon, Portugal

REFERENCES:
- [Result] Silva AM, Armada-da-Silva P, Sardinha LB, Júdice PB, Magalhães JP, Matias CN & Santos DA. Efeitos da ingestão de cafeína na água corporal total, distribuição de fluidos intra e extracelulares e no dispêndio energético. A Report for the Institution of Hydration and Health, In press.
- [Result] Júdice PB (2011). Determinant Factors on hydration status assessed by Urine Specific Gravity: accuracy of technical procedures and effect of caffeine ingestion. Master's Degree Thesis. Faculty of Human Kinetics-Technical University of Lisbon, Cruz-Quebrada.
- [Result] Magalhães JP, Santos DA, Silva AM, Matias CN, Júdice PB, Quintas IC, Sardinha LB (2011). Total energy expenditure: combined heart rate and motion sensor vs uni-axial accelerometry models Book of abstracts of the International conference on Recent Advances and Controversies in Measuring Energy Metabolism, pp 106.
- [Result] Quintas IC, Santos DA, Matias CN, Silva AM, Gobbo, LA, Gonçalves EM, Magalhães JP, Júdice PB, Sardinha LB (2011). Does caffeine intake affect resting energy expenditure? Book of abstracts of the International conference on Recent Advances and Controversies in Measuring Energy Metabolism, pp 104.
- [Result] Júdice PB, Silva AM, Magalhães JP, Matias CN, Santos DA, Armada-da-Silva P, & Sardinha LB. Does caffeine intake increases energy expenditure and habitual physical activity? A double-blind randomized crossover trial. Medicine and Science in Sports and Exercise. In Review.
- [Derived] Francisco R, Rosa GB, Judice PB, Magalhaes JP, Cruz AD, Sardinha LB, Lukaski HC, Silva AM. Four days of a moderate dose of caffeine does not alter raw bioelectrical impedance analysis parameters in healthy males. Clin Nutr ESPEN. 2025 Oct;69:599-607. doi: 10.1016/j.clnesp.2025.08.005. Epub 2025 Aug 6. PMID 40774622
- [Derived] Silva AM, Santos DA, Matias CN, Judice PB, Magalhaes JP, Ekelund U, Sardinha LB. Accuracy of a combined heart rate and motion sensor for assessing energy expenditure in free-living adults during a double-blind crossover caffeine trial using doubly labeled water as the reference method. Eur J Clin Nutr. 2015 Jan;69(1):20-7. doi: 10.1038/ejcn.2014.51. Epub 2014 Apr 2. PMID 24690589
- [Derived] Judice PB, Matias CN, Santos DA, Magalhaes JP, Hamilton MT, Sardinha LB, Silva AM. Caffeine intake, short bouts of physical activity, and energy expenditure: a double-blind randomized crossover trial. PLoS One. 2013 Jul 15;8(7):e68936. doi: 10.1371/journal.pone.0068936. Print 2013. PMID 23869233
- [Derived] Silva AM, Judice PB, Matias CN, Santos DA, Magalhaes JP, St-Onge MP, Goncalves EM, Armada-da-Silva P, Sardinha LB. Total body water and its compartments are not affected by ingesting a moderate dose of caffeine in healthy young adult males. Appl Physiol Nutr Metab. 2013 Jun;38(6):626-32. doi: 10.1139/apnm-2012-0253. Epub 2013 Jan 15. PMID 23724879
- [Derived] Judice PB, Magalhaes JP, Santos DA, Matias CN, Carita AI, Armada-Da-Silva PA, Sardinha LB, Silva AM. A moderate dose of caffeine ingestion does not change energy expenditure but decreases sleep time in physically active males: a double-blind randomized controlled trial. Appl Physiol Nutr Metab. 2013 Jan;38(1):49-56. doi: 10.1139/apnm-2012-0145. Epub 2013 Jan 18. PMID 23368828